CLINICAL TRIAL: NCT05898581
Title: Ultrasound-guided Pericapsular Nerve Group (PENG) Block vs. Intraoperative Local Anesthetic Infiltration (ILAI) for Total Hip Arthroplasty (THA): a Single Center, Non-inferiority Randomized Control Trial Pilot Study.
Brief Title: PENG Block vs. Intraoperative Local Anesthetic Infiltration for Total Hip Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, MD, Anesthesiologist, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PENG RCT
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Anesthesia
Keywords: anesthesia; total hip arthroplasty; Pericapsular Nerve Group Block
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study will be a single-centre, double-blinded non-inferiority randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG Block (Experimental): Participants will receive ultrasound-guided PENG block (PENG group) with local anesthetics (20 ml of 0.5% ropivacaine) before administration of spinal anesthesia. Patients in this group will also receive a sham ILAI procedure with 60 mL of saline (performed by the operating surgeon).
  Interventions: Procedure: PENG Block
- Control Group (Sham Comparator): Participants will receive a sham PENG block performed with 20ml of normal saline solution before spinal anesthesia. After, patients will receive ILAI (performed by the operating surgeon) with a plain solution of ropivacaine 0.25% 60ml.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: PENG Block — Participants will receive a PENG block with local anesthetics (which is a freezing medication, in this case, 0.5% ropivacaine) before receiving spinal anesthesia. Patients in this group will also receive a sham ILAI procedure with 60 mL of saline (performed by the operating surgeon).
  Arms: PENG Block
Procedure: Control Group — Participants will receive a sham PENG block performed with 20ml of normal saline solution before spinal anesthesia. After, patients will receive ILAI (performed by the operating surgeon) with a plain solution of ropivacaine 0.25% 60ml.
  Arms: Control Group

SUMMARY:
Currently, the analgesic standard of care for patients undergoing total hip arthroplasty (THA) at our centre is intraoperative infiltration with a solution of local anesthetic, morphine (opioid), and ketorolac (nonsteroidal anti-inflammatory drug - NSAID). If a patient has a contraindication for the use of an opioid or NSAIDs, this infiltration is performed with a plain local anesthetic. No blocks (numbing of certain nerves to prevent pain from occurring in that area) are performed for postoperative pain in these patients. The pericapsular nerve group (PENG) block is a recently described technique with limited data in the literature that has assessed the benefits of using this nerve block for THA procedures. The purpose of this study is to investigate if the ultrasound-guided PENG block can provide non-inferior postoperative analgesia compared to local intraoperative anesthetic infiltration (ILAI) with an associated cost benefit for patients undergoing THA.

DETAILED DESCRIPTION:
Traditionally, the most common ultrasound-guided nerve blocks utilized for hip analgesia during THA are the Femoral Nerve Block and the Fascia Iliaca Block. Despite the analgesia component of both techniques, they can cause quadriceps weakness1-2, which is an unwanted side effect for this patient population as it interferes with surgical recovery, physical therapy, and increases the risk of fall. For these reasons, these types of blocks are not performed for patients undergoing THA at our center (London Health Science Centre).

In 2018, a cadaveric study performed by Short et al. demonstrated that the hip capsule is innervated by sensory branches of the Femoral Nerve and Accessory Obturator Nerves.3 An ultrasound-guided technique for the blockade of the articular branches of the hip was first described by Giron-Arango et al.4 The major benefit of using this approach is the possible motor-sparing effect, capable of maintaining the quadriceps muscle force as the technique aims only at sensory articular branches.

The current standard care for postoperative analgesia for THA is intraoperative infiltration with a solution containing ropivacaine 0.25% (local anesthetic), morphine (opioid), and ketorolac (NSAID). Patients with any contra-indication for the administration of opioids, or nonsteroidal anti-inflammatories receive intraoperative infiltration with plain local anesthetic.

The efficacy of ILAI for THA remains inconclusive. While some studies validated the benefit of this technique5-9, others were not able to confirm improvements in pain control.10-15 As it is a simple technique based on the injection of analgesic solution in the tissue surrounding the surgical field, it has become a popular intervention.

Similarly, the analgesic efficacy of the PENG block for THA remains unclear. As the PENG block involves sensory articular nerves of the anterior hip capsule, the benefit for the patients lies in the possibility of having a good analgesic response along with no motor leg weakness. This will improve patient care during the postoperative period with early mobilization and adequate pain control. There is limited information in the literature available regarding the use of the PENG block as part of the postoperative analgesia plan for THA. Thus, we have identified a need to conduct a trial that aims to investigate if the ultrasound-guided PENG block can provide non-inferior postoperative analgesia compared to local intraoperative anesthetic infiltration (ILAI).

In 2020, a retrospective case series by Kukreja et al16 evaluated twelve patients that underwent total hip arthroplasty (six primaries, six revisions). This study showed a decrease in opioid consumption in the primary THA group. In this group, two patients had spinal anesthesia as the primary anesthesia technique, while four received general anesthetic. Hence, the results of this study have suggested that the PENG block may be useful for postoperative analgesia in this procedure.

Following this case report series, Aliste et al17 conducted a randomized trial comparing the ultrasound-guided PENG block with the ultrasound-guided suprainguinal fascia iliaca block with the purpose of evaluating the postoperative incidence of quadriceps motor block as the primary outcome. In this study, the PENG block resulted in a lower incidence of quadriceps motor block compared with the suprainguinal fascia iliaca block.

In addition, two randomized clinical trials were conducted in 2022 involving the addition of the ultrasound-guided PENG block in the analgesic plan for patients that underwent THA demonstrating benefits. Both of these studies demonstrated benefits of incorporating the PENG block into the analgesic care plan for this patient population. First, Lin et al18 conducted a randomized clinical trial in which patients received either a PENG block or a sham block in addition to spinal anesthesia and ILAI (100ml of ropivacaine 0.1% with 1mg of epinephrine). In this study, the patients that received the PENG block had less postoperative pain with preservation of quadriceps muscle strength.

Second, Zheng et al19 performed a similar randomized trial in which patients undergoing THA were randomized to the intervention group that received the PENG block, or to the placebo group in which a PENG block was simulated with an injection of 20ml of normal saline solution. All patients had general anesthesia as the main anesthetic plan and received an ILAI with 20ml of ropivacaine 0.5% by the end of the procedure. The study showed that the addition of a PENG block provided a limited advantage to postoperative analgesia in the Post-Anesthesia Care Unit (PACU) and lower intraoperative opioid consumption.

At this point, in our understanding, no further clinical data is available comparing the analgesic efficacy of PENG block with ILAI. Further clinical trials are needed to test the efficacy of PENG blocks.

Following consent, patients will be randomized to one of two study groups (on a 1:1 basis):

Group 1: patients will receive ultrasound-guided PENG block (PENG group) with local anesthetics (20 ml of 0.5% ropivacaine) before administration of spinal anesthesia. Patients in this group will also receive a sham ILAI procedure with 60 mL of saline (performed by the operating surgeon).

Group 2: patients will receive a sham PENG block performed with 20ml of normal saline solution before spinal anesthesia. After, patients will receive ILAI (performed by the operating surgeon) with a plain solution of ropivacaine 0.25% 60ml.

The block group (PENG group), will be administered a single dose of ultrasound-guided PENG block with 20ml of ropivacaine 0.5% drawn up by an anesthesiologist in the BR before the spinal anesthesia. All patients will be offered Midazolam 1-2 mg IV before the start of the interventions. In the control group, a sham PENG block with 20ml of normal saline will be performed before spinal anesthesia. After, ILAI will be performed by the operating surgeon with a plain solution of ropivacaine 0.25% 60ml. In both groups, the anesthesiologist will be blinded to perform the PENG and Sham block. Next, spinal anesthesia will be performed with bupivacaine 0.5% 15mg intrathecally. The spinal anesthesia will be tested for sensory block to cold using an alcoholic chlorhexidine pad, and for motor block by asking the patient to move either leg. The timing of the completion of the spinal anesthesia will be marked and it will be considered time zero. Next, the patient will be moved to the main OR for surgery. Intraoperative sedation will be at the discretion of the OR anesthesiologist. If spinal anesthesia fails, the patient will receive general anesthetic in the operating room. This patient will however remain in the study group as "intention to treat".

A blinded data collector will record all outcomes (NRS pain score, PACU length, muscle strength, and intraoperative opioid consumption). The timing of the completion of the spinal anesthesia will be considered time zero. At 8 hours and 24 hours after the end of the spinal anesthesia, the patient will be approached by the blinded data assessor to collect the NRS pain score. Pain score evaluation will be recorded at rest, on passive movement, and on active movement of the operated hip joint. Also, the quadriceps muscle strength will be evaluated by the capacity of the patient to perform knee extension at 8 hours and 24 hours postoperatively. Data will be collected for the patient's opioid consumption in the 24 hours after the spinal anesthesia was completed. Pain assessment and muscle strength will be evaluated using the following scales:

Pain assessment: A Likert-like numerical rating scale (NRS) will be used for pain assessment, 0 = no pain, 1-3= mild pain, 4-6= moderate pain interfering with activity, and 7-10= severe, disabling pain.

Muscle strength: The quadriceps muscle function will be evaluated. Strength testing of the quadriceps will include the resistance of knee extension and hip flexion. Commonly used muscle testing grading will be used:

Grade 5: Full range of motion against gravity with maximal resistance Grade 4: Full range of motion against gravity, moderate resistance Grade 3: Full range of motion against gravity Grade 2: Full range of motion, gravity eliminated Grade 1: Visible or palpable contraction without motion Grade 0: No visible or palpable contraction

All patients will be offered oral opioids on an as-needed basis. The total amount of opioids administered to the patient in the 24 hours after the neuraxial procedure will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (>18 years old)
2. Undergoing THA with a direct lateral surgical approach (transgluteal approach)
3. Ability to provide verbal/written consent to participate in this trial

Exclusion Criteria:

1. Patient with any contraindication for spinal anesthesia
2. Patient with any contraindication for regional analgesia
3. Patient undergoing THA with a direct anterior surgical approach
4. Patients undergoing THA for hip revision
5. Patients undergoing THA under One Day Stay (ODS) admission
6. Patients that received opioids intrathecally
7. Patients having residual motor block six hours after the completion of the spinal anesthesia.
8. Patients with a history of regular opioid intake for more than three months
9. Patients incapable of performing knee extension of the same operative side
10. Pregnant patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
PENG block impact on post-operative pain scores | 8-24 hours following completion of spinal anesthesia
  Patient pain scores will be evaluated at 8 hours and 24 hours following completion of spinal anesthesia to determine the impact of the PENG block on post-operative pain. Pain scores will be assessed using a Likert scale rating (0-10, 0 = no pain, 10 = sever, disabling pain).

SECONDARY OUTCOMES:
PENG block impact on quadriceps muscle strength post-operatively | 8-24 hours following completion of spinal anesthesia
  Patient's quadricep strength will be evaluated at 8 hours and 24 hours following completion of spinal anesthesia to determine the impact of the PENG block on quadricep muscle strength. This will be evaluated by assessing the ability of the patient to perform knee extensions and hip flexion. Muscle strength grading will be evaluated using the following grading system:
  Grade 5: Full range of motion against gravity with maximal resistance Grade 4: Full range of motion against gravity, moderate resistance Grade 3: Full range of motion against gravity Grade 2: Full range of motion, gravity eliminated Grade 1: Visible or palpable contraction without motion Grade 0: No visible or palpable contraction
Time spent in post-anesthesia care unit (PACU) following surgery | Up to 24 hours following completion of spinal anesthesia.
  The time patient's spend in the PACU following surgery will be evaluated to determine if the administration of the PENG block has any impact on this outcome. This will be measured by recording the time the patient entered and exited the PACU.
Patient opioid consumption 24 hours period after spinal anesthesia procedure. | 24 hours following following completion of spinal anesthesia.
  Amount of opioids that were consumed by the patient following surgery. This is being evaluated to determine if administration of the PENG block has any impact on this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, FRCPC, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behrends M, Yap EN, Zhang AL, Kolodzie K, Kinjo S, Harbell MW, Aleshi P. Preoperative Fascia Iliaca Block Does Not Improve Analgesia after Arthroscopic Hip Surgery, but Causes Quadriceps Muscles Weakness: A Randomized, Double-blind Trial. Anesthesiology. 2018 Sep;129(3):536-543. doi: 10.1097/ALN.0000000000002321. PMID 29975203
- [Background] Xing JG, Abdallah FW, Brull R, Oldfield S, Dold A, Murnaghan ML, Whelan DB. Preoperative Femoral Nerve Block for Hip Arthroscopy: A Randomized, Triple-Masked Controlled Trial. Am J Sports Med. 2015 Nov;43(11):2680-7. doi: 10.1177/0363546515602468. Epub 2015 Sep 24. PMID 26403206
- [Background] Short AJ, Barnett JJG, Gofeld M, Baig E, Lam K, Agur AMR, Peng PWH. Anatomic Study of Innervation of the Anterior Hip Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 Feb;43(2):186-192. doi: 10.1097/AAP.0000000000000701. PMID 29140962
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Ban WR, Zhang EA, Lv LF, Dang XQ, Zhang C. Effects of periarticular injection on analgesic effects and NSAID use in total knee arthroplasty and total hip arthroplasty. Clinics (Sao Paulo). 2017 Dec;72(12):729-736. doi: 10.6061/clinics/2017(12)03. PMID 29319718
- [Background] Villatte G, Engels E, Erivan R, Mulliez A, Caumon N, Boisgard S, Descamps S. Effect of local anaesthetic wound infiltration on acute pain and bleeding after primary total hip arthroplasty: the EDIPO randomised controlled study. Int Orthop. 2016 Nov;40(11):2255-2260. doi: 10.1007/s00264-016-3133-3. Epub 2016 Feb 22. PMID 26899484
- [Background] Murphy TP, Byrne DP, Curtin P, Baker JF, Mulhall KJ. Can a periarticular levobupivacaine injection reduce postoperative opiate consumption during primary hip arthroplasty? Clin Orthop Relat Res. 2012 Apr;470(4):1151-7. doi: 10.1007/s11999-011-2108-3. Epub 2011 Sep 30. PMID 21960156
- [Background] Liu W, Cong R, Li X, Wu Y, Wu H. Reduced opioid consumption and improved early rehabilitation with local and intraarticular cocktail analgesic injection in total hip arthroplasty: a randomized controlled clinical trial. Pain Med. 2011 Mar;12(3):387-93. doi: 10.1111/j.1526-4637.2010.01043.x. Epub 2011 Jan 25. PMID 21266004
- [Background] Busch CA, Whitehouse MR, Shore BJ, MacDonald SJ, McCalden RW, Bourne RB. The efficacy of periarticular multimodal drug infiltration in total hip arthroplasty. Clin Orthop Relat Res. 2010 Aug;468(8):2152-9. doi: 10.1007/s11999-009-1198-7. Epub 2009 Dec 18. PMID 20020333
- [Background] Hofstad JK, Winther SB, Rian T, Foss OA, Husby OS, Wik TS. Perioperative local infiltration anesthesia with ropivacaine has no effect on postoperative pain after total hip arthroplasty. Acta Orthop. 2015;86(6):654-8. doi: 10.3109/17453674.2015.1053775. Epub 2015 May 22. PMID 25997827
- [Background] den Hartog YM, Mathijssen NM, van Dasselaar NT, Langendijk PN, Vehmeijer SB. No effect of the infiltration of local anaesthetic for total hip arthroplasty using an anterior approach: a randomised placebo controlled trial. Bone Joint J. 2015 Jun;97-B(6):734-40. doi: 10.1302/0301-620X.97B6.35343. PMID 26033051
- [Background] Zoric L, Cuvillon P, Alonso S, Demattei C, Vialles N, Asencio G, Ripart J, Nouvellon E. Single-shot intraoperative local anaesthetic infiltration does not reduce morphine consumption after total hip arthroplasty: a double-blinded placebo-controlled randomized study. Br J Anaesth. 2014 Apr;112(4):722-8. doi: 10.1093/bja/aet439. Epub 2014 Jan 14. PMID 24431385
- [Background] Lunn TH, Husted H, Solgaard S, Kristensen BB, Otte KS, Kjersgaard AG, Gaarn-Larsen L, Kehlet H. Intraoperative local infiltration analgesia for early analgesia after total hip arthroplasty: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2011 Sep-Oct;36(5):424-9. doi: 10.1097/AAP.0b013e3182186866. PMID 21610559
- [Background] Hirasawa N, Kurosaka K, Nishino M, Nakayama T, Matsubara M, Tsukada S. No Clinically Important Difference in Pain Scores After THA Between Periarticular Analgesic Injection and Placebo: A Randomized Trial. Clin Orthop Relat Res. 2018 Sep;476(9):1837-1845. doi: 10.1097/CORR.0000000000000374. PMID 29939894
- [Background] Dobie I, Bennett D, Spence DJ, Murray JM, Beverland DE. Periarticular local anesthesia does not improve pain or mobility after THA. Clin Orthop Relat Res. 2012 Jul;470(7):1958-65. doi: 10.1007/s11999-012-2241-7. Epub 2012 Jan 24. PMID 22270468
- [Background] Kukreja P, Avila A, Northern T, Dangle J, Kolli S, Kalagara H. A Retrospective Case Series of Pericapsular Nerve Group (PENG) Block for Primary Versus Revision Total Hip Arthroplasty Analgesia. Cureus. 2020 May 19;12(5):e8200. doi: 10.7759/cureus.8200. PMID 32572357
- [Background] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085
- [Background] Lin DY, Brown B, Morrison C, Fraser NS, Chooi CSL, Cehic MG, McLeod DH, Henningsen MD, Sladojevic N, Kroon HM, Jaarsma RL. The Pericapsular Nerve Group (PENG) block combined with Local Infiltration Analgesia (LIA) compared to placebo and LIA in hip arthroplasty surgery: a multi-center double-blinded randomized-controlled trial. BMC Anesthesiol. 2022 Aug 6;22(1):252. doi: 10.1186/s12871-022-01787-2. PMID 35933328
- [Background] Zheng J, Pan D, Zheng B, Ruan X. Preoperative pericapsular nerve group (PENG) block for total hip arthroplasty: a randomized, placebo-controlled trial. Reg Anesth Pain Med. 2022 Mar;47(3):155-160. doi: 10.1136/rapm-2021-103228. Epub 2021 Dec 6. PMID 34873023
- See also: Joint replacement at LHSC — https://www.lhsc.on.ca/joint-replacement-surgery